CLINICAL TRIAL: NCT07273864
Title: A Randomized Controlled Trial of Auricular Thumbtack Needle Therapy Combined With Conventional Treatment and Median Nerve Electrical Stimulation on Consciousness Recovery Prognosis and Family Satisfaction in Craniocerebral Injury Patients With Consciousness Disorder
Brief Title: Effect of Median Nerve Electrical Stimulation Combined With Auricular Acupuncture on Consciousness Disturbance in Patients With Craniocerebral Injury
Acronym: ANECT-CCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Li Hai (Other)
Responsible Party: Sponsor-Investigator, Li Hai, Chief Therapist, Department of Rehabilitation, First Affiliated Hospital of Gannan Medical University
Organization: First Affiliated Hospital of Gannan Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LLSL-2022053105
Record Dates: First submitted 2025-10-01; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Traumatic Brain Injury; Cerebral Hemorrhage
Keywords: Traumatic Brain Injury; Median Nerve Electrical Stimulation; Disorders of Consciousness; Promotion of Arousal; Ear Acupoint Press-Needl
MeSH Terms: conditions — Brain Injuries, Traumatic; Cerebral Hemorrhage; Consciousness Disorders | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Treatment + Median Nerve Electrical Stimulation + Auricular Press-Needle Therapy (Experimental): Conventional treatment combined with right median nerve electrical stimulation and auricular press-needle therapy.
  Interventions: Other: Conventional Neurosurgical and Supportive Care; Device: Right Median Nerve Electrical Stimulation; Device: Auricular Press-Needle Therapy
- Conventional Treatment + Median Nerve Electrical Stimulation (Active Comparator): Conventional treatment combined with right median nerve electrical stimulation.
  Interventions: Other: Conventional Neurosurgical and Supportive Care; Device: Right Median Nerve Electrical Stimulation

INTERVENTIONS:
Other: Conventional Neurosurgical and Supportive Care — Routine comprehensive management for severe traumatic brain injury, including surgical intervention when indicated, intracranial pressure monitoring if needed, neuroprotective and symptomatic medications (e.g., anti-epileptic drugs), nutritional support, complication prevention, nursing care, and conventional rehabilitation therapy. All care was provided in accordance with institutional standard protocols.
Device: Right Median Nerve Electrical Stimulation — The multifunctional electrical therapy apparatus (Model MT1023; Shenzhen Dongdixin Technology Co., Ltd.) was used. A single skin electrode was placed 2 cm proximal to the right wrist crease on the volar forearm. Stimulation parameters: asymmetric biphasic (direct current) square wave, intensity up to 20 mA, pulse width 300 ms, frequency 40 Hz, intermittent mode (20 seconds on, 40 seconds off). Sessions lasted 60 minutes and were delivered twice daily, 7 days per week, for 8 weeks.
Device: Auricular Press-Needle Therapy — Disposable sterile press needles (0.2 mm × 0.5 mm thumbtack type) were inserted bilaterally at the auricular acupoints Shenmen (TF4) and Subcortex/Brain (AT4) [some records also included Heart (CO15) and Sympathetic]. Needles were retained for 48 hours, replaced every 2-3 days, and the cycle was repeated for the entire 8-week treatment period. Family members were trained to massage each point three times daily.
  Arms: Conventional Treatment + Median Nerve Electrical Stimulation + Auricular Press-Needle Therapy

SUMMARY:
This study aims to evaluate the effects of auricular press needle therapy, combined with conventional treatment and median nerve electrical stimulation, on promoting arousal and neurological recovery in patients with disorders of consciousness after traumatic brain injury.

Sixty patients with a Glasgow Coma Scale (GCS) score of 4-8 were enrolled and randomly assigned in a 1:1 ratio to a control group or an experimental group (30 patients each). Both groups received standard conventional treatment (including surgery when indicated, medications, nutritional support, acupuncture, and complication prevention) combined with median nerve electrical stimulation. The experimental group received auricular press needle therapy (at Heart, Shenmen, Sympathetic, and Subcortex acupoints) on top of the same interventions, and family members were trained to perform daily acupoint massage.

The GCS score and Coma Recovery Scale-Revised (CRS-R) score were assessed at baseline, 4 weeks, 6 weeks, and 8 weeks after the start of intervention, and the arousal rate was recorded. The Glasgow Outcome Scale (GOS) was used to evaluate prognosis at 1 month after the end of treatment, and family satisfaction was assessed using a Likert scale at 8 weeks post-intervention. Data were analyzed using SPSS Statistics 27.0, with statistical significance set at p < 0.05.

DETAILED DESCRIPTION:
This was a single-center, parallel-group, randomized controlled trial. Patients were stratified by injury severity according to the Glasgow Coma Scale (GCS 4-6 versus 7-8) and randomized 1:1 using a computer-generated sequence produced by an independent statistician.

Allocation was concealed with sequentially numbered opaque sealed envelopes opened only after informed consent had been signed by legal guardians.

Blinding of patients, families, and therapists was not feasible due to the visible auricular needles and stimulation device. Outcome assessors remained blinded throughout; they received uniform training, used scoring forms without intervention information, and were regularly supervised.

Both groups received conventional treatment (surgery when indicated, medication, nutritional support, acupuncture, and complication prevention) plus right median nerve electrical stimulation twice daily for 8 weeks (40 Hz, 300 ms pulse width, intensity gradually increased to 20 mA). The experimental group additionally received auricular press needle therapy at Heart, Shenmen, Sympathetic, and Subcortex acupoints (disposable sterile needles, 3 days on/1 day off cycle, repeated throughout the 8 weeks), with family members trained to massage the points three times daily for 10 minutes.

All staff completed standardized training and passed competency checks. Weekly supervision by a senior neurosurgeon ensured treatment fidelity, data integrity, and family compliance.

Outcome assessments were conducted within 24 hours of enrollment (baseline: demographics, Glasgow Coma Scale [GCS], Coma Recovery Scale-Revised [CRS-R], duration of consciousness disturbance, imaging findings, and vital signs), at 4 and 6 weeks (awakening status, GCS, CRS-R, adverse events, and treatment compliance), at 8 weeks (awakening rate, GCS, CRS-R, and family satisfaction), and at 12 weeks (1 month after completion of the 8-week intervention: Glasgow Outcome Scale [GOS] for long-term prognosis).

Data were recorded on standardized electronic case report forms with double-entry by two independent clerks. Discrepancies were resolved by referring to original records and the supervisor. The database was password-protected, accessible only to authorized personnel, and backed up weekly both on-site and off-site.

Safety was monitored daily and adverse events were graded and managed according to a predefined protocol. Sample size of 60 patients (30 per group) was calculated to detect an increase in 8-week awakening rate from 40 % to 70 % (α=0.05, two-sided; power=0.80; 10 % dropout).

Statistical analyses were performed using SPSS 27.0 and R 4.2.1. All tests were two-sided with statistical significance set at p < 0.05. The primary outcome (8-week awakening rate) was analyzed with the χ² test. Secondary outcomes were analyzed using repeated-measures ANOVA for GCS/CRS-R scores, Kaplan-Meier and log-rank test for time-to-awakening, Mann-Whitney U test or ordinal regression for GOS, and t-test/χ² test for family satisfaction. Both intention-to-treat (ITT) and per-protocol (PP) analyses were conducted as sensitivity analyses. Pre-specified subgroup analyses were performed according to initial injury severity (GCS 4-6 versus 7-8) and duration of consciousness disturbance before enrollment (< 5 days versus 5-10 days).

ELIGIBILITY:
Inclusion Criteria:

* Disorder of consciousness following traumatic brain injury
* Stable vital signs with no evidence of active bleeding
* Glasgow Coma Scale (GCS) score between 4 and 8 (inclusive)
* No severe vital organ dysfunction and normal cardiac function
* Time from injury to enrollment ≤ 10 days
* No prior history of traumatic brain injury, epilepsy, or pregnancy

Exclusion Criteria:

* Presence of other critical illnesses (e.g., severe cardiovascular, hepatic, or renal disease)
* Known allergy to the electrodes or adhesive patches used in electrical stimulation
* Lack of cooperation or refusal by the patient's legal guardian/family members

Ages: 20 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Awakening Rate of Patients with Consciousness Disorder After Traumatic Brain Injury (TBI) | 8 weeks after the start of the intervention (which is the end of the full intervention course for the study).
  1. Description Primary outcome is awakening rate at 8 weeks post-intervention in TBI patients with consciousness disorder (GCS 4-8). "Awakening" = independent eye-opening ≥30s, or clear responses (limb retraction, simple verbal answers) to verbal/pain stimuli, confirmed by 2 attending physicians.
  2. Time Frame 8 weeks after intervention start (end of full course).
  3. Assessment Method Record weekly awakening status during 8-week intervention; Count awakened patients in Arm 1 (control) and Arm 2 (experimental) at week 8; Calculate rate: (Awakened patients / Total patients per group) × 100%.
  4. Rationale Awakening is core rehabilitation goal for these patients, directly reflecting intervention efficacy in consciousness recovery. More intuitive and clinically meaningful than other indicators (e.g., GCS) for evaluating core therapeutic effect.

SECONDARY OUTCOMES:
Change in Glasgow Coma Scale (GCS) Score | Baseline (pre-intervention), 4 weeks, 6 weeks, 8 weeks post-intervention.
  Description: Change in GCS score (3-15 points; higher = better neurofunction) from baseline to 4, 6, 8 weeks post-intervention.
  Time Frame: Baseline (pre-intervention), 4 weeks, 6 weeks, 8 weeks post-intervention.
  Method: Trained nurses assess GCS (eye-opening, verbal, motor responses); calculate score changes (post-intervention - baseline).
  Rationale: Supplements awakening rate, quantifies gradual neurofunctional improvement over intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Hai N Li, Middle Initia, Study Chair — First Affiliated Hospital of Gannan Medical University
Locations (1):
- The First Affiliated Hospital of Gannan Medical University, Jiangxi, Ganzhou, China

IPD SHARING:
Plan to Share IPD: No
Patient Privacy Protection:
  Collected IPD includes sensitive personal health information. Per China's Personal Information Protection Law and hospital ethical requirements, sharing IPD risks unauthorized disclosure, violating patients' information security rights.
  Informed Consent Limitations :
  Participants' signed consent only authorizes IPD use for this study's research goals, not sharing with external parties. Without additional ethical approval and patient re-consent, sharing is non-compliant with ethical commitments.
  Data Security & Integrity :
  IPD is managed under The First Affiliated Hospital of Gannan Medical University's security system. External sharing may cause data tampering, improper use, or loss, compromising result integrity and analysis credibility.
  Future IPD sharing (e.g., collaborative research) will require hospital Ethics Committee approval, patient re-consent, and strict de-identification/transfer protocols to meet legal and ethical standards.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-30): https://cdn.clinicaltrials.gov/large-docs/64/NCT07273864/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT07273864/ICF_001.pdf